CLINICAL TRIAL: NCT03828877
Title: The Effect of Acupuncture on Pain, IL 17 and IL 23 in Endovenous Ablation; Prospective, Randomized, Controlled Study.
Brief Title: The Effect of Acupuncture on the Treatment of Endovenous Ablation on Pain, IL17 and IL 23
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Yavuz Orak, Assistant Professor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2018/13-26
Record Dates: First submitted 2019-01-29; First posted 2019-02-04 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Pain; Interleukin; Vessels; Varicose
Keywords: Acupuncture, Pain , IL 17, IL 23 and Vessel
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group C (No Intervention): Arm: Group C control group. Non-acupuncture group. Gruop C will be Control group.
- Group A (Active Comparator): Arm: Group A, group of acupuncture Akupunktur will be done with Pres Needle (0.22x1.5 mm) Blood will be taken for the measurement of IL 17 and IL 23 from Group A (Acupuncture) patients 24 hours prior to endovenous ablation procedure. Then, with press needle (0.22x1.5) LU 9 (Taiyuan), LU7 (Lieque), SP 6 (Sanyinjiao) , ST 36 (Zusanli), LI 4 (Hegu) and LIV 3 (Taichong) points will be applied acupuncture.On the 3rd day, patients will be called for control. Blood will also be taken from the blood to measure IL 17, IL 23 values.
  Interventions: Other: Group A ( Group Acupuncture)

INTERVENTIONS:
Other: Group A ( Group Acupuncture) — Group A; Acupunctur will be done with Pres Needle (0.22x1.5 mm).Acupuncture will be done points fo SP 6, LI 4 , ST 36 , LİV 3, LU 9 ,LU 7.
  Arms: Group A

SUMMARY:
Acupuncture has emerged in China about 2,000 years ago and is one of the oldest medical procedures in the world. Acupuncture continued to evolve and develop over the centuries, and gradually became one of the standard treatments used in China. Introduced to other regions such as Asia, Europe and the United States. The most extensive use of acupuncture is for pain relief. The aim of this study was to prevent complications due to pain frequently seen in patients who would be treated with endovenous ablation in the postoperative period. In addition, the effect of acupuncture on operative hemodynamics, pain, vascular diameter, postoperative, nausea, vomiting, pain and analgesic needs, IL17 and IL 23.

DETAILED DESCRIPTION:
Patients will be divided into two groups. Control group (Group C, n: 35) and Acupuncture group (Group A, n: 35). Inclusion criteria: willing to participate in the study, being in the 18-65 age range, a saphenous vein diameter greater than 5.5 mm and a small saphenous vein diameter of less than 4 mm with reflux for greater than 0.5 s The patients with the study will be taken.Exclusion criteria: patients outside the 18-65 age range, patients with deep venous system obstruction, patients who have previously used another invasive treatment method (thermal and chemical ablation, surgery), patients with heart and kidney failure, patients with secondary varicose veins patients with hypercoagulable state, patients with local or systemic infection, patients with obesity (body mass index> 35), patients with impaired consciousness, patients who do not want to participate in the study. Blood will be taken from Group A and Group C patients for the measurement of IL 17 and IL 23 prior 24 hours before the endovenous ablation procedure. Group A will be done LU 9 (Taiyuan), LU 7 (Lieque), SP 6 (Sanyinjiao) , ST 36 (Suzanli), LI 4 (Hegu) and LIV 3 (Taichong) points to be acupunctured. Vasculer access will be opened in the preoperative patient preparation room in both patient groups.The points of the acupuncture group will be checked and recorded. The falling press needle will be reapplied to replace the needles. Patients will be taken to the operating room. In both patient groups, measurement of the vessel diameter by ultrasound before the endovenous ablation procedure will be performed.During the endovenous ablation procedure, SBP (Systolic blood pressure), DBP (Diastolic blood pressure), OAB (Mean arterial pressure), HR (Heart rate), SPO2 (Oxygen) , the number of interventional procedures needed to be successful and the duration of the procedure, the pain conditions during operation (VAS) will be recorded in 1, 3, 5, 7, 10, 15 minutes.After completion of the procedure, ultrasound vein ablation and measurement will be reassessed by the surgeon to evaluate the success of the procedure.Nausea, vomiting, itching and pain conditions (VAS) will be measured again in the postoperative 1, 30 and 60 minutes and a comparison will be made between the groups.After the operation, the acupuncture points will be checked in the postoperative resting room and if there are falling needles, the needles will be replaced again.Patients will be told that acupuncture points should be stimulated from time to time and pres needle needles should be protected for three days.On the 3rd postoperative day, patients will be referred to the cardiovascular surgery outpatient clinic. Pain conditions (VAS) and analgesic consumption will be evaluated.Preoperatively, postoperatively and on the 3rd day, the vessel diameters will be measured and compared with ultrasonography.IL17 and IL 23 values will be compared between both groups and before and after endovenous ablation.The effect of acupuncture on IL 17 and IL 23 will be investigated.Patients will also be told to return to the hospital immediately in cases such as shortness of breath, edema, redness, pain in the legs and the complications will be recorded.The aim of this study was to investigate the effect of acupuncture on pain, IL17, IL 23 and vessel diameters in patients treated with N-Butyl Cyanoacrylate, a new method in the treatment of endovenous ablation.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers to participate in the study,
* 18-65 years of age,
* patients with a saphenous vein diameter greater than 5.5 mm
* small saphenous vein diameter of less than 4 mm with reflux for greater than 0.5 s

Exclusion Criteria:

* Patients outside the 18-65 age range,
* patients with deep venous system obstruction,
* patients who have previously used another invasive treatment method (thermal and chemical ablation, surgery),
* patients with heart and kidney failure,
* patients with secondary varicose veins,
* patients with hypercoagulable state patients,
* patients with local or systemic infections,
* patients with obesity (body mass index> 35),
* patients with impaired consciousness,
* patients who do not want to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2019-03-05 (Actual); Study Completion 2019-03-07 (Actual)

PRIMARY OUTCOMES:
IL 17 and IL 23 values | before operation and after the operation 3. days
  Change From Baseline on the circulating levels of IL 17 and IL 23 ng/ L
Pain (VAS Score) | Change From Baseline of VAS Score in 1 minute,3 minute,5 minute,7 minute, 10 minute, 15 minute of pain level during operation.Each unit will be evaluated separately within itself
  Change from Baseline VAS Score. from 1 to 10 , 0: No pain, 10: 10 pain that can not be tolerated
Pain (VAS Score) | Change From Baseline of VAS Score in1 minute,30 minute, 60 minute after operation and 3. days. Each unit will be evaluated separately within itself
  Change from Baseline VAS Score (Visual analog scale) Score. from 1 to 10 , 0: No pain, 10: 10 pain that can not be tolerated

SECONDARY OUTCOMES:
vessel measurement | before the operation, after operation and after operation 3. days
  Change from Baseline measurement (mm)with ultrasonografi

CONTACTS AND LOCATIONS:
Overall Officials: yavuz orak, Principal Investigator — Kahramanmaraş Sutcu Imam University Faculty of Medicine Kahramanmaraş
Locations (1):
- Kahramanmaras Sutcu Imam University Faculty of Medicine, Kahramanmaraş, Onikişubat, Turkey (Türkiye)